CLINICAL TRIAL: NCT02339155
Title: A Randomized, Open-label Study to Evaluate the Immunogenicity of Anthrax Vaccine Adsorbed Alone or Concomitantly With Raxibacumab (GSK3068483)
Brief Title: Effect of Raxibacumab on Immunogenicity of Anthrax Vaccine Adsorbed
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emergent BioSolutions (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201436
Record Dates: First submitted 2015-01-12; First posted 2015-01-15 (Estimated); Results first posted 2018-01-09 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Infections, Bacterial
Keywords: Anthrax Vaccine Adsorbed; Raxibacumab; Immunogenicity
MeSH Terms: conditions — Bacterial Infections | interventions — raxibacumab; Diphenhydramine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anthrax Vaccine Adsorbed (Experimental): Subjects will be administered subcutaneous (SC) 0.5 mL AVA doses on Days 1, 15, and 29 (0, 2, and 4 weeks).
  Interventions: Biological: AVA
- AVA + Raxibacumab (Experimental): Subjects will be administered SC 0.5 mL AVA doses on Days 1, 15, and 29 (0, 2, and 4 weeks), with the first AVA dose administered immediately after completion of a single intravenous (IV) infusion 40 milligram (mg)/kilogram (kg) raxibacumab dose. Subjects will be premedicated with 25-50 mg of diphenhydramine up to 1 hour prior to the raxibacumab infusion to reduce the risk of infusion reactions.
  Interventions: Biological: AVA; Biological: Raxibacumab; Drug: Diphenhydramine

INTERVENTIONS:
Biological: AVA — Sterile, milky-white suspension with dosage level of 0.5 mL for SC administration
Biological: Raxibacumab — Sterile, liquid formulation with unit dose strength of 40 mg/ kg for IV administration
  Arms: AVA + Raxibacumab
Drug: Diphenhydramine — Depending upon the labelling of the specific product chosen, 25 - 50 mg will be administered orally or IV
  Arms: AVA + Raxibacumab

SUMMARY:
This study, as a post-marketing commitment to the Food and Drug Administration, is designed to detect the effect of raxibacumab on anthrax vaccine adsorbed (AVA) immunogenicity in a healthy volunteer population. This is a randomized, open-label, parallel group, two arm study to compare the immunogenicity of AVA at 4 weeks after the first AVA dose, when AVA is administered alone or concomitantly with raxibacumab. The study is planned to enroll approximately 30 to 534 subjects in up to 3 cohorts. The total duration of the study will be approximately 26 weeks. The dates reflect cohort 1.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by the Investigator or medically qualified designee based on a medical evaluation including medical history, physical examination and laboratory tests
* Men and women between 18 to 65 years of age
* Willing and able to adhere to the procedures stated in the protocol.
* Female subject is eligible to participate if she is not pregnant (as confirmed by a negative serum or urine human chorionic gonadotrophin (hCG) test), not lactating, and at least one of the following conditions applies:

Non-reproductive potential defined as:

Pre-menopausal females with one of the following: Documented tubal ligation, Documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion, Hysterectomy, Documented Bilateral Oophorectomy Postmenopausal defined as 12 months of spontaneous amenorrhea. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment.

Reproductive potential and agrees to follow one of the options listed in the GSK Modified List of Highly Effective Methods for Avoiding Pregnancy in Females of Reproductive Potential (FRP), from 30 days prior to the first dose of study medication and until after the last dose of study medication and completion of the follow-up visit at Day 183 (at least five terminal half-lives for raxibacumab).

Exclusion Criteria:

* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or non-investigational study vaccine/product (pharmaceutical product or device).
* Be a member of the military, a laboratory worker, first responder, health care worker, or otherwise be at higher risk of exposure to anthrax.
* History of regular alcohol consumption within 1 month of the study defined as:

An average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 g of alcohol: 12 ounces (360 milliliter [mL]) of beer, 5 ounces (150 mL) of wine or 1.5 ounces (45 mL) of 80 proof distilled spirits.

* Female planning to become pregnant or planning to discontinue contraceptive precautions before the Day 183 study visit.
* Pregnant (confirmed by a serum or urine hCG test) or lactating female.
* Alanine aminotransferase (ALT) and bilirubin >1.5 x upper limit of normal (ULN) (isolated bilirubin >1.5 x ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Any confirmed or suspected immunosuppressive or immunodeficient condition resulting from disease (e.g., malignancy, human immunodeficiency virus [HIV] infection) or immunosuppressive/cytotoxic therapy (e.g., medications used during cancer chemotherapy, organ transplantation or to treat autoimmune disorders).
* Presence of hepatitis B surface antigen (HBsAg), positive hepatitis C antibody test results at screening or within 3 months prior to first dose of study treatment.
* A positive pre-study drug/alcohol screen.
* A positive test for HIV antibody.
* History of sensitivity to any of the study medications, or components thereof (especially latex and aluminium) or a history of other known drug allergies that, in the opinion of the Investigator or GSK Medical Monitor, contraindicates their participation.
* Have previously been vaccinated against PA.
* Have an anti-PA Ab concentration >2 times the lower limit of quantitation at screening.
* Administration of immunoglobulins not included in this trial and/or any blood products within the 3 months preceding the first dose of study vaccine or planned administration during the study period.
* Administration of long-acting immune-modifying drugs (e.g. infliximab) within six months prior to the first vaccine dose or expected administration at any time during the study period.
* Chronic administration (defined as more than 14 consecutive days) of systemic immunosupressants or other immune-modifying drugs within six months prior to the first vaccine dose. Inhaled, topical and intra-articular corticosteroids are allowed.
* Administration or planned administration of a vaccine not foreseen by the study protocol within the period starting 35 days before the first dose of study vaccine(s) and ending 30 days after the last dose of study vaccine. This includes any type of vaccine such as (but not limited to) live, inactivated, and subunit vaccines. Influenza vaccines are permitted after Week 8.
* Subjects must abstain from taking prescription or non-prescription drugs (including vitamins and dietary or herbal supplements), within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication until completion of the follow-up visit, unless in the opinion of the Investigator and sponsor the medication will not interfere with the study.
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Any condition which, in the opinion of the investigator, prevents the subject from participating in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 573 (Actual)
Dates: Start 2015-02-24 (Actual); Primary Completion 2017-01-03 (Actual); Study Completion 2017-06-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul-Andre deLame, MD, Study Director — Emergent BioSolutions Inc
Locations (3):
- United States (3):
  - GSK Investigational Site, Edgewater, Florida
  - GSK Investigational Site, Overland Park, Kansas
  - GSK Investigational Site, Knoxville, Tennessee

REFERENCES:
- [Derived] Skoura N, Wang-Jairaj J, Della Pasqua O, Chandrasekaran V, Billiard J, Yeakey A, Smith W, Steel H, Tan LK. Effect of raxibacumab on immunogenicity of Anthrax Vaccine Adsorbed: a phase 4, open-label, parallel-group, randomised non-inferiority study. Lancet Infect Dis. 2020 Aug;20(8):983-991. doi: 10.1016/S1473-3099(20)30069-4. Epub 2020 Apr 22. PMID 32333847

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study included healthy volunteers who were not previously immunized against protective antigen. 573 participants were randomized with 566 receiving study treatment and 537 completed the study.
Pre-assignment Details: A total of 573 participants were randomized with 566 receiving study treatment and 537 completed the study.
Groups:
- AVA Alone: Participants administered Anthrax vaccine adsorbed (AVA) subcutaneous (SC) 0.5 milliliter (mL) on Days 1, 15 and 29
- AVA+Raxibacumab: Participants administered SC 0.5 mL of AVA doses on Days 1, 15, and 29. with the first AVA dose administered immediately after completion of a single 40 milligram/kilogram (mg/kg) intravenous (IV) infusion of raxibacumab dose (Day 1). Participants were premedicated with 25-50 mg of diphenhydramine up to 1 hour prior to the raxibacumab infusion to reduce the risk of infusion reactions.
Period: Overall Study
Arm/Group | AVA Alone | AVA+Raxibacumab
Started (This includes Intent-to-treat population (ITT)) | 287 | 286
Received Study Treatment | 286 | 280
Completed | 272 | 265
Not Completed | 15 | 21
Not completed — Adverse Event | 0 | 6
Not completed — Death | 1 | 1
Not completed — Lost to Follow-up | 8 | 9
Not completed — Physician Decision | 2 | 1
Not completed — Withdrawal by Subject | 4 | 4

BASELINE CHARACTERISTICS:
Population: The Intent to Treat (ITT) Population comprised of all randomized participants
Groups:
- AVA Alone: Participants administered AVA SC, 0.5 mL on Days 1, 15 and 29
- AVA+Raxibacumab: Participants administered SC 0.5 mL of AVA doses on Days 1, 15, and 29, with the first AVA dose administered immediately after completion of a single 40 mg/kg, IV infusion of raxibacumab dose (Day 1). Participants were premedicated with 25-50 mg of diphenhydramine up to 1 hour prior to the raxibacumab infusion to reduce the risk of infusion reactions.
- Total: Total of all reporting groups
Arm/Group | AVA Alone | AVA+Raxibacumab | Total
Number analyzed (Participants) | 287 | 286 | 573
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: The ITT Population comprised of all randomized participants
  Years | 36.2 (12.78) | 36.1 (12.06) | 36.2 (12.42)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: ITT
  Participants
    Female | 150 | 142 | 292
    Male | 137 | 144 | 281
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: ITT
  Participants
    White | 216 | 221 | 437
    Black or African American | 61 | 56 | 117
    American Indian or Alaska Native | 7 | 1 | 8
    Asian | 2 | 5 | 7
    Multiple | 1 | 2 | 3
    Unknown | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Ratio of Geometric Mean Concentrations (GMC) of Anti-protective Antigen (PA) Antibody (Ab) at 4 Weeks (Day 29) After the First AVA Dose (Prior to the Third AVA Dose), Between the AVA Alone and the AVA With Raxibacumab Treatment Groups
Description: Ratio of the GMC of anti-PA Ab between AVA alone and the AVA with raxibacumab treatment group was assessed to compare the immunogenicity of AVA at 4 weeks after the first AVA dose (prior to the third AVA dose). Serum AVA derived anti-PA Ab concentrations were determined using an approved immunoassay. Per Protocol (PP) population was used in analysis which comprised of all analyzable participants (those who received at least the Week 0 [Day 1] and Week 2 [Day 15] AVA doses within the protocol specified visit window; receive the raxibacumab dose, if randomized to Treatment Group 2 and; completed the primary study endpoint assessment [anti-PA Ab concentration at Week 4]).
Time Frame: Day 29
Population: PP Population.
Measure: Geometric Mean (95% Confidence Interval); unit: Microgram/milliliter (µg/mL)
Arm/Group | AVA Alone | AVA+Raxibacumab
Number analyzed (Participants) | 276 | 269
Microgram/milliliter (µg/mL) | 26.516 [23.580 to 29.816] | 22.477 [20.098 to 25.137]
Statistical Analysis 1: Comparison: AVA Alone vs AVA+Raxibacumab; Test type: Non-Inferiority — If the upper bound of the 90% confidence interval (CI) or the ratio of anti-PA Ab (attributable to AVA) GMCs between the AVA and the AVA + raxibacumab groups at Week 4 is less than 1.5, non-inferiority was to be established; p = 0.0016, t-test, 1 sided; Ratio = 1.18, 90% CI 2-sided [1.03 to 1.35]

2. Secondary Outcome: Ratio of GMC of Anti-PA Ab at Weeks 8 and 26 (Days 57 and 183) After the First AVA Dose, Between the AVA Alone and AVA With Raxibacumab Treatment Groups
Description: Anti-PA antibody concentrations were collected at Weeks 8 and 26 after the first AVA dose. Serum AVA derived anti-PA Ab concentrations were determined using an approved immunoassay. The GMCs with corresponding 95% CI were calculated for each treatment group at each timepoint. Only those participants available at the specified time points (represented by n=X in the category titles) were analyzed.
Time Frame: Days 57 and 183
Population: PP Population.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | AVA Alone | AVA+Raxibacumab
Number analyzed (Participants) | 275 | 267
µg/mL
  Week 8, n=275, 267 | 50.470 [46.124 to 55.224] | 46.095 [41.860 to 50.757]
  Week 26, n=267, 258: number analyzed (Participants) | 267 | 258
  Week 26, n=267, 258 | 10.007 [9.243 to 10.835] | 10.231 [9.479 to 11.042]
Statistical Analysis 1: Comparison: AVA Alone vs AVA+Raxibacumab; Test type: Other; t-test, 1 sided; Ratio = 1.09, 90% CI 2-sided [0.98 to 1.22] — Week 8
Statistical Analysis 2: Comparison: AVA Alone vs AVA+Raxibacumab; Test type: Other; p < 0.0001, t-test, 1 sided; Ratio = 0.98, 90% CI 2-sided [0.89 to 1.07] — Week 26

3. Secondary Outcome: Percentage of Participants Who Seroconvert, at Weeks 4, 8, and 26 (Days 29, 57 and 183) After the First AVA Dose, Between the AVA Alone and the AVA With Raxibacumab Treatment Groups
Description: The percentage of participants, with corresponding 95% CI based on Wilson's method, who seroconvert (seroconversion is defined as a >4-fold increase in toxin neutralizing activity [TNA] titer) was summarized, at Weeks 4, 8 and 26 after the first AVA dose for both arms separately. Serum TNA titer was determined using a cell-based assay.
Time Frame: Days 29, 57 and 183
Population: PP Population.
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | AVA Alone | AVA+Raxibacumab
Number analyzed (Participants) | 276 | 269
Percent of Participants
  Week 4 | 76.4 [71.1 to 81.1] | 99.3 [97.3 to 99.8]
  Week 8 | 95.3 [92.5 to 97.5] | 98.1 [96.7 to 99.6]
  Week 26 | 31.9 [27.6 to 38.8] | 32.0 [27.9 to 39.3]

4. Secondary Outcome: Number of Participants With Any Serious Adverse Event (SAE) and Any Non-serious Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE resulting in death, is life threatening (ie, an immediate threat to life), inpatient hospitalization, prolongation of existing hospitalization, persistent or significant disability/incapacity, congenital anomaly/birth defect or any other situation which is medically important and may jeopardize the participant or may require medical or surgical intervention or events associated with liver injury and impaired liver function is categorized as SAE. The Safety population was comprised of all randomized participants who received at least one dose of AVA.
Time Frame: Up to Day 183
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | AVA Alone | AVA+Raxibacumab
Number analyzed (Participants) | 286 | 280
Participants
  Non-serious AEs | 85 | 80
  SAE | 5 | 3

5. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) at Indicated Time Points
Description: SBP and DBP were measured in semi-supine position after 5 minutes rest. Values at Day -1 were considered as Baseline values. Change from Baseline was defined as difference between the post-Baseline visit value and the Baseline value. Only those participants available at the specified time points (represented by n=X in the category titles) were analyzed.
Time Frame: Baseline and up to Day 183
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Millimeter of mercury (mmHg)
Groups:
- AVA+Raxibacumab: Participants administered SC 0.5 mL of AVA doses on Days 1, 15, and 29. with the first AVA dose administered immediately after completion of a single 40 mg/kg, IV infusion of raxibacumab dose (Day 1). Participants were premedicated with 25-50 mg of diphenhydramine up to 1 hour prior to the raxibacumab infusion to reduce the risk of infusion reactions.
Arm/Group | AVA Alone | AVA+Raxibacumab
Number analyzed (Participants) | 286 | 280
Millimeter of mercury (mmHg)
  SBP, Day 1, n=286, 280 | -3.4 (9.2) | -3.8 (9.6)
  SBP, Day 29, n=283, 279: number analyzed (Participants) | 283 | 279
  SBP, Day 29, n=283, 279 | 0.6 (9.9) | 1.9 (9.9)
  SBP, Day 57, n=282, 275: number analyzed (Participants) | 282 | 275
  SBP, Day 57, n=282, 275 | 1.8 (10.9) | 2.2 (10.3)
  SBP, Day 183, n=273, 266: number analyzed (Participants) | 273 | 266
  SBP, Day 183, n=273, 266 | 2.4 (10.6) | 1.5 (9.9)
  DBP, Day 1, n=286, 280 | -2.7 (6.9) | -3.1 (6.8)
  DBP, Day 29, n=283, 279: number analyzed (Participants) | 283 | 279
  DBP, Day 29, n=283, 279 | 1.0 (7.3) | 1.6 (6.5)
  DBP, Day 57, n=282, 275: number analyzed (Participants) | 282 | 275
  DBP, Day 57, n=282, 275 | 1.9 (7.4) | 2.3 (7.4)
  DBP, Day 183, n=273, 266: number analyzed (Participants) | 273 | 266
  DBP, Day 183, n=273, 266 | 2.3 (8.4) | 2.5 (7.9)

6. Secondary Outcome: Change From Baseline in Heart Rate at Indicated Time Points
Description: Heart rate was measured in semi-supine position after 5 minutes rest. Values at Day -1 were considered as Baseline values. Change from Baseline was defined as difference between the post-Baseline visit value and the Baseline value. Only those participants available at the specified time points (represented by n=X in the category titles) were analyzed.
Time Frame: Baseline and up to Day 183
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Beats per minute (bpm)
Arm/Group | AVA Alone | AVA+Raxibacumab
Number analyzed (Participants) | 286 | 280
Beats per minute (bpm)
  Day 1, n=286, 280 | -0.3 (10.4) | -0.8 (10.5)
  Day 29, n=283, 279: number analyzed (Participants) | 283 | 279
  Day 29, n=283, 279 | -0.4 (10.5) | -0.4 (10.5)
  Day 57, n=282, 275: number analyzed (Participants) | 282 | 275
  Day 57, n=282, 275 | -1.2 (10.6) | -0.9 (11.2)
  Day 183, n=273, 266: number analyzed (Participants) | 273 | 266
  Day 183, n=273, 266 | 0.9 (11.7) | 0.7 (11.5)

7. Secondary Outcome: Change From Baseline in Respiratory Rate at Indicated Time Points
Description: Respiratory rate was measured in semi-supine position after 5 minutes rest. Values at Day -1 were considered as Baseline values. Change from Baseline was defined as difference between the post-Baseline visit value and the Baseline value. Only those participants available at the specified time points (represented by n=X in the category titles) were analyzed.
Time Frame: Baseline and up to Day 183
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | AVA Alone | AVA+Raxibacumab
Number analyzed (Participants) | 286 | 280
Breaths per minute
  Day 1, n=286, 280 | -0.4 (1.5) | -0.3 (1.5)
  Day 29, n=283, 279: number analyzed (Participants) | 283 | 279
  Day 29, n=283, 279 | -0.1 (1.4) | -0.1 (1.4)
  Day 57, n=282, 276: number analyzed (Participants) | 282 | 276
  Day 57, n=282, 276 | -0.1 (1.5) | -0.1 (1.3)
  Day 183, n=273, 266: number analyzed (Participants) | 273 | 266
  Day 183, n=273, 266 | -0.3 (1.6) | -0.2 (1.5)

8. Secondary Outcome: Change From Baseline in Temperature at Indicated Time Points
Description: Temperature was measured in semi-supine position after 5 minutes rest. Values at Day -1 were considered as Baseline values. Change from Baseline was defined as difference between the post-Baseline visit value and the Baseline value. Only those participants available at the specified time points (represented by n=X in the category titles) were analyzed.
Time Frame: Baseline and up to Day 183
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Degree celsius
Arm/Group | AVA Alone | AVA+Raxibacumab
Number analyzed (Participants) | 286 | 280
Degree celsius
  Day 1, n=286, 280 | -0.04 (0.26) | 0.02 (0.27)
  Day 29, n=283, 279: number analyzed (Participants) | 283 | 279
  Day 29, n=283, 279 | -0.04 (0.24) | -0.03 (0.31)
  Day 57, n=282, 276: number analyzed (Participants) | 282 | 276
  Day 57, n=282, 276 | -0.05 (0.25) | -0.02 (0.25)
  Day 183, n=272, 266: number analyzed (Participants) | 272 | 266
  Day 183, n=272, 266 | -0.04 (0.277) | -0.01 (0.26)

9. Secondary Outcome: Number of Participants With Hematology Parameters Outside Normal Range
Description: Hematology parameters included assessment of platelet count, erythrocytes, leukocytes , reticulocyte count, mean corpuscular volume (MCV), mean corpuscular hemoglobin (MCH), mean corpuscular hemoglobin concentration (MCHC), neutrophils, lymphocytes, monocytes, eosinophils, basophils, hemoglobin and hematocrit. Here high is equal to above the upper limit of the normal range, low is equal to below the lower limit of the normal range. Participants are counted in the category that their value changes to (low, normal or high), unless there is no change in their category. Only those participants available at the specified time points (represented by n=X in the category titles) were analyzed.
Time Frame: Up to Day 57
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | AVA Alone | AVA+Raxibacumab
Number analyzed (Participants) | 286 | 280
Participants
  Eosinophils 10^9/Liter (L) Low, Week 4, n=282, 278: number analyzed (Participants) | 282 | 278
  Eosinophils 10^9/Liter (L) Low, Week 4, n=282, 278 | 0 | 0
  Eosinophils 10^9/L High, Week 4, n=282, 278: number analyzed (Participants) | 282 | 278
  Eosinophils 10^9/L High, Week 4, n=282, 278 | 4 | 6
  Eosinophils 10^9/L, Low, Week 8, n=281, 276: number analyzed (Participants) | 281 | 276
  Eosinophils 10^9/L, Low, Week 8, n=281, 276 | 0 | 0
  Eosinophils 10^9/L, High, Week 8, n=281, 276: number analyzed (Participants) | 281 | 276
  Eosinophils 10^9/L, High, Week 8, n=281, 276 | 7 | 5
  Basophils 10^9/L, Low, Week 4, n=282, 278: number analyzed (Participants) | 282 | 278
  Basophils 10^9/L, Low, Week 4, n=282, 278 | 0 | 0
  Basophils 10^9/L, High, Week 4, n=282, 278: number analyzed (Participants) | 282 | 278
  Basophils 10^9/L, High, Week 4, n=282, 278 | 0 | 0
  Basophils 10^9/L, Low, Week 8, n=281, 276: number analyzed (Participants) | 281 | 276
  Basophils 10^9/L, Low, Week 8, n=281, 276 | 0 | 0
  Basophils 10^9/L, High, Week 8, n=281, 276: number analyzed (Participants) | 281 | 276
  Basophils 10^9/L, High, Week 8, n=281, 276 | 0 | 0
  Hematocrit percent (%) Low, Week 4, n=283, 279: number analyzed (Participants) | 283 | 279
  Hematocrit percent (%) Low, Week 4, n=283, 279 | 7 | 6
  Hematocrit %, High, Week 4, n=283, 279: number analyzed (Participants) | 283 | 279
  Hematocrit %, High, Week 4, n=283, 279 | 2 | 1
  Hematocrit %, Low, Week 8, n=281, 276: number analyzed (Participants) | 281 | 276
  Hematocrit %, Low, Week 8, n=281, 276 | 6 | 9
  Hematocrit %, High, Week 8, n=281, 276: number analyzed (Participants) | 281 | 276
  Hematocrit %, High, Week 8, n=281, 276 | 2 | 2
  Hemoglobin gram/Liter (g/L) Low,Week 4,n=283, 279: number analyzed (Participants) | 283 | 279
  Hemoglobin gram/Liter (g/L) Low,Week 4,n=283, 279 | 7 | 3
  Hemoglobin g/L, High, Week 4, n=283, 279: number analyzed (Participants) | 283 | 279
  Hemoglobin g/L, High, Week 4, n=283, 279 | 4 | 1
  Hemoglobin g/L, Low, Week 8, n=281, 276: number analyzed (Participants) | 281 | 276
  Hemoglobin g/L, Low, Week 8, n=281, 276 | 7 | 10
  Hemoglobin g/L, High, Week 8, n=281, 276: number analyzed (Participants) | 281 | 276
  Hemoglobin g/L, High, Week 8, n=281, 276 | 3 | 2
  Lymphocytes 10^9/L , Low, Week 4, n=282, 278: number analyzed (Participants) | 282 | 278
  Lymphocytes 10^9/L , Low, Week 4, n=282, 278 | 3 | 1
  Lymphocytes 10^9/L , High, Week 4, n=282, 278: number analyzed (Participants) | 282 | 278
  Lymphocytes 10^9/L , High, Week 4, n=282, 278 | 0 | 1
  Lymphocytes 10^9/L, Low, Week 8, n=281, 276: number analyzed (Participants) | 281 | 276
  Lymphocytes 10^9/L, Low, Week 8, n=281, 276 | 2 | 4
  Lymphocytes 10^9/L, High, Week 8, n=281, 276: number analyzed (Participants) | 281 | 276
  Lymphocytes 10^9/L, High, Week 8, n=281, 276 | 0 | 0
  MCH picogram (pg), Low, Week 4, n=283, 279: number analyzed (Participants) | 283 | 279
  MCH picogram (pg), Low, Week 4, n=283, 279 | 2 | 1
  MCH pg, High, Week 4, n=283, 279: number analyzed (Participants) | 283 | 279
  MCH pg, High, Week 4, n=283, 279 | 0 | 0
  MCH pg, Low, Week 8, n=281, 276: number analyzed (Participants) | 281 | 276
  MCH pg, Low, Week 8, n=281, 276 | 2 | 5
  MCH pg, High, Week 8, n=281, 276: number analyzed (Participants) | 281 | 276
  MCH pg, High, Week 8, n=281, 276 | 0 | 0
  MCHC g/L, Low, Week 4, n=283, 279: number analyzed (Participants) | 283 | 279
  MCHC g/L, Low, Week 4, n=283, 279 | 3 | 3
  MCHC g/L, High, Week 4, n=283, 279: number analyzed (Participants) | 283 | 279
  MCHC g/L, High, Week 4, n=283, 279 | 19 | 17
  MCHC g/L, Low, Week 8, n=281, 276: number analyzed (Participants) | 281 | 276
  MCHC g/L, Low, Week 8, n=281, 276 | 3 | 7
  MCHC g/L, High, Week 8, n=281, 276: number analyzed (Participants) | 281 | 276
  MCHC g/L, High, Week 8, n=281, 276 | 16 | 12
  MCV femtoliters (fL), Low, Week 4, n=283, 279: number analyzed (Participants) | 283 | 279
  MCV femtoliters (fL), Low, Week 4, n=283, 279 | 2 | 2
  MCV fL, High, Week 4, n=283, 279: number analyzed (Participants) | 283 | 279
  MCV fL, High, Week 4, n=283, 279 | 0 | 1
  MCV fL, Low, Week 8, n=281, 276: number analyzed (Participants) | 281 | 276
  MCV fL, Low, Week 8, n=281, 276 | 3 | 2
  MCV fL, High, Week 8, n=281, 276: number analyzed (Participants) | 281 | 276
  MCV fL, High, Week 8, n=281, 276 | 0 | 0
  Monocytes 10^9/L , Low, Week 4, n=282, 278: number analyzed (Participants) | 282 | 278
  Monocytes 10^9/L , Low, Week 4, n=282, 278 | 0 | 0
  Monocytes 10^9/L, High, Week 4, n=282, 278: number analyzed (Participants) | 282 | 278
  Monocytes 10^9/L, High, Week 4, n=282, 278 | 3 | 2
  Monocytes 10^9/L, Low, Week 8, n=281, 276: number analyzed (Participants) | 281 | 276
  Monocytes 10^9/L, Low, Week 8, n=281, 276 | 0 | 0
  Monocytes 10^9/L, High, Week 8, n=281, 276: number analyzed (Participants) | 281 | 276
  Monocytes 10^9/L, High, Week 8, n=281, 276 | 0 | 1
  Neutrophils 10^9/L, Low, Week 4, n=283, 279: number analyzed (Participants) | 283 | 279
  Neutrophils 10^9/L, Low, Week 4, n=283, 279 | 7 | 8
  Neutrophils 10^9/L, High, Week 4, n=283, 279: number analyzed (Participants) | 283 | 279
  Neutrophils 10^9/L, High, Week 4, n=283, 279 | 3 | 2
  Neutrophils 10^9/L, Low, Week 8, n=281, 276: number analyzed (Participants) | 281 | 276
  Neutrophils 10^9/L, Low, Week 8, n=281, 276 | 5 | 6
  Neutrophils 10^9/L, High, Week 8, n=281, 276: number analyzed (Participants) | 281 | 276
  Neutrophils 10^9/L, High, Week 8, n=281, 276 | 1 | 6
  Erythrocytes 10^12/L, Low, Week 4, n=283, 279: number analyzed (Participants) | 283 | 279
  Erythrocytes 10^12/L, Low, Week 4, n=283, 279 | 6 | 4
  Erythrocytes 10^12/L, High, Week 4, n=283, 279: number analyzed (Participants) | 283 | 279
  Erythrocytes 10^12/L, High, Week 4, n=283, 279 | 4 | 7
  Erythrocytes 10^12/L, Low, Week 8, n=281, 276: number analyzed (Participants) | 281 | 276
  Erythrocytes 10^12/L, Low, Week 8, n=281, 276 | 2 | 8
  Erythrocytes 10^12/L, High, Week 8, n=281, 276: number analyzed (Participants) | 281 | 276
  Erythrocytes 10^12/L, High, Week 8, n=281, 276 | 6 | 3
  Leukocytes 10^9/L, Low, Week 4, n=283, 279: number analyzed (Participants) | 283 | 279
  Leukocytes 10^9/L, Low, Week 4, n=283, 279 | 15 | 12
  Leukocytes 10^9/L, High, Week 4, n=283, 279: number analyzed (Participants) | 283 | 279
  Leukocytes 10^9/L, High, Week 4, n=283, 279 | 2 | 2
  Leukocytes 10^9/L, Low, Week 8, n=281, 276: number analyzed (Participants) | 281 | 276
  Leukocytes 10^9/L, Low, Week 8, n=281, 276 | 6 | 10
  Leukocytes 10^9/L, High, Week 8, n=281, 276: number analyzed (Participants) | 281 | 276
  Leukocytes 10^9/L, High, Week 8, n=281, 276 | 1 | 5
  Reticulocytes 10^12/L, Low, Week 4, n=283, 279: number analyzed (Participants) | 283 | 279
  Reticulocytes 10^12/L, Low, Week 4, n=283, 279 | 1 | 0
  Reticulocytes 10^12/L, High, Week 4, n=283, 279: number analyzed (Participants) | 283 | 279
  Reticulocytes 10^12/L, High, Week 4, n=283, 279 | 1 | 3
  Reticulocytes 10^12/L, Low, Week 8, n=281, 276: number analyzed (Participants) | 281 | 276
  Reticulocytes 10^12/L, Low, Week 8, n=281, 276 | 1 | 1
  Reticulocytes 10^12/L, High, Week 8, n=281, 276: number analyzed (Participants) | 281 | 276
  Reticulocytes 10^12/L, High, Week 8, n=281, 276 | 5 | 3
  Platelet 10^9/L, Low, Week 4, n=282, 279: number analyzed (Participants) | 282 | 279
  Platelet 10^9/L, Low, Week 4, n=282, 279 | 6 | 4
  Platelet 10^9/L, High, Week 4, n=282, 279: number analyzed (Participants) | 282 | 279
  Platelet 10^9/L, High, Week 4, n=282, 279 | 0 | 0
  Platelet 10^9/L, Low, Week 8, n=280, 276: number analyzed (Participants) | 280 | 276
  Platelet 10^9/L, Low, Week 8, n=280, 276 | 4 | 4
  Platelet 10^9/L, High, Week 8, n=280, 276: number analyzed (Participants) | 280 | 276
  Platelet 10^9/L, High, Week 8, n=280, 276 | 1 | 0

10. Secondary Outcome: Number of Participants With Clinical Chemistry Parameters Outside Normal Range
Description: Blood samples were collected to evaluate clinical chemistry parameters, which included assessment of urea nitrogen (UN), creatinine, chloride, glucose, magnesium, total protein, potassium, chloride, total Carbon dioxide (CO2), sodium, calcium (cal), alkaline phosphatase (ALP), aspartate aminotransferase (AST), alanine aminotransferase (ALT), gamma-glutamyltransferase (GGT), total and direct bilirubin ( D.bili), albumin and calculated creatinine clearance. Here high is equal to above the upper limit of the normal range, low is equal to below the lower limit of the normal range. Participants are counted in the category that their value changes to (low, normal or high), unless there is no change in their category. Only those participants available at the specified time points (represented by n=X in the category titles) were analyzed.
Time Frame: Up to Day 57
Population: Safety Population.
Measure: Number; unit: Participants
Arm/Group | AVA Alone | AVA+Raxibacumab
Number analyzed (Participants) | 286 | 280
Participants
  Albumin g/L, Low, Week 4, n=283, 279: number analyzed (Participants) | 283 | 279
  Albumin g/L, Low, Week 4, n=283, 279 | 6 | 2
  Albumin g/L, High, Week 4, n=283, 279: number analyzed (Participants) | 283 | 279
  Albumin g/L, High, Week 4, n=283, 279 | 1 | 0
  Albumin g/L, Low, Week 8, n=282, 275: number analyzed (Participants) | 282 | 275
  Albumin g/L, Low, Week 8, n=282, 275 | 2 | 1
  Albumin g/L, High, Week 8, n=282, 275: number analyzed (Participants) | 282 | 275
  Albumin g/L, High, Week 8, n=282, 275 | 0 | 0
  ALP units/liter (U/L), Low, Week 4, n=283, 279: number analyzed (Participants) | 283 | 279
  ALP units/liter (U/L), Low, Week 4, n=283, 279 | 3 | 5
  ALP U/L, High, Week 4, n=283, 279: number analyzed (Participants) | 283 | 279
  ALP U/L, High, Week 4, n=283, 279 | 14 | 20
  ALP U/L, Low, Week 8, n=282, 275: number analyzed (Participants) | 282 | 275
  ALP U/L, Low, Week 8, n=282, 275 | 2 | 2
  ALP U/L, High, Week 8, n=282, 275: number analyzed (Participants) | 282 | 275
  ALP U/L, High, Week 8, n=282, 275 | 13 | 19
  ALT U/L, Low, Week 4, n=283, 279: number analyzed (Participants) | 283 | 279
  ALT U/L, Low, Week 4, n=283, 279 | 45 | 44
  ALT U/L, High, Week 4, n=283, 279: number analyzed (Participants) | 283 | 279
  ALT U/L, High, Week 4, n=283, 279 | 7 | 4
  ALT U/L, Low, Week 8, n=282, 275: number analyzed (Participants) | 282 | 275
  ALT U/L, Low, Week 8, n=282, 275 | 39 | 42
  ALT U/L, High, Week 8, n=282, 275: number analyzed (Participants) | 282 | 275
  ALT U/L, High, Week 8, n=282, 275 | 7 | 6
  AST U/L, Low, Week 4, n=283, 279: number analyzed (Participants) | 283 | 279
  AST U/L, Low, Week 4, n=283, 279 | 41 | 37
  AST U/L, High, Week 4, n=283, 279: number analyzed (Participants) | 283 | 279
  AST U/L, High, Week 4, n=283, 279 | 7 | 5
  AST U/L, Low, Week 8, n=282, 275: number analyzed (Participants) | 282 | 275
  AST U/L, Low, Week 8, n=282, 275 | 38 | 34
  AST U/L, High, Week 8, n=282, 275: number analyzed (Participants) | 282 | 275
  AST U/L, High, Week 8, n=282, 275 | 6 | 10
  D.bili micromole/Liter (µmol/L) LowWeek4,n=274,263: number analyzed (Participants) | 274 | 263
  D.bili micromole/Liter (µmol/L) LowWeek4,n=274,263 | 0 | 0
  D.bili µmol/L, High, Week 4, n=274, 263: number analyzed (Participants) | 274 | 263
  D.bili µmol/L, High, Week 4, n=274, 263 | 5 | 3
  D.bili µmol/L, Low, Week 8, n=274, 261: number analyzed (Participants) | 274 | 261
  D.bili µmol/L, Low, Week 8, n=274, 261 | 0 | 0
  D.bili µmol/L, High, Week 8, n=274, 261: number analyzed (Participants) | 274 | 261
  D.bili µmol/L, High, Week 8, n=274, 261 | 5 | 9
  Bili µmol/L, Low, Week 4, n=280, 279: number analyzed (Participants) | 280 | 279
  Bili µmol/L, Low, Week 4, n=280, 279 | 5 | 4
  Bili µmol/L, High, Week 4, n=280, 279: number analyzed (Participants) | 280 | 279
  Bili µmol/L, High, Week 4, n=280, 279 | 1 | 5
  Bili µmol/L, Low, Week 8, n=280, 273: number analyzed (Participants) | 280 | 273
  Bili µmol/L, Low, Week 8, n=280, 273 | 3 | 2
  Bili µmol/L, High, Week 8, n=280, 273: number analyzed (Participants) | 280 | 273
  Bili µmol/L, High, Week 8, n=280, 273 | 2 | 7
  Cal,millimole/Liter (mmol/L)Low,Week 4,n=283, 279: number analyzed (Participants) | 283 | 279
  Cal,millimole/Liter (mmol/L)Low,Week 4,n=283, 279 | 6 | 4
  Cal mmol/L, High, Week 4, n=283, 279: number analyzed (Participants) | 283 | 279
  Cal mmol/L, High, Week 4, n=283, 279 | 2 | 4
  Cal mmol/L, Low, Week 8, n=282, 275: number analyzed (Participants) | 282 | 275
  Cal mmol/L, Low, Week 8, n=282, 275 | 12 | 10
  Cal mmol/L, High, Week 8, n=282, 275: number analyzed (Participants) | 282 | 275
  Cal mmol/L, High, Week 8, n=282, 275 | 0 | 3
  Chloride mmol/L, Low, Week 4, n=283, 279: number analyzed (Participants) | 283 | 279
  Chloride mmol/L, Low, Week 4, n=283, 279 | 0 | 0
  Chloride mmol/L, High, Week 4, n=283, 279: number analyzed (Participants) | 283 | 279
  Chloride mmol/L, High, Week 4, n=283, 279 | 19 | 12
  Chloride mmol/L, Low, Week 8, n=282, 275: number analyzed (Participants) | 282 | 275
  Chloride mmol/L, Low, Week 8, n=282, 275 | 0 | 0
  Chloride mmol/L, High, Week 8, n=282, 275: number analyzed (Participants) | 282 | 275
  Chloride mmol/L, High, Week 8, n=282, 275 | 12 | 9
  CO2 mmol/L, Low, Week 4, n=283, 279: number analyzed (Participants) | 283 | 279
  CO2 mmol/L, Low, Week 4, n=283, 279 | 7 | 11
  CO2 mmol/L, High, Week 4, n=283, 279: number analyzed (Participants) | 283 | 279
  CO2 mmol/L, High, Week 4, n=283, 279 | 14 | 12
  CO2 mmol/L, Low, Week 8, n=282, 275: number analyzed (Participants) | 282 | 275
  CO2 mmol/L, Low, Week 8, n=282, 275 | 6 | 14
  CO2 mmol/L, High, Week 8, n=282, 275: number analyzed (Participants) | 282 | 275
  CO2 mmol/L, High, Week 8, n=282, 275 | 10 | 9
  Creatinine µmol/L, Low, Week 4, n=283, 279: number analyzed (Participants) | 283 | 279
  Creatinine µmol/L, Low, Week 4, n=283, 279 | 19 | 10
  Creatinine µmol/L, High, Week 4, n=283, 279: number analyzed (Participants) | 283 | 279
  Creatinine µmol/L, High, Week 4, n=283, 279 | 6 | 3
  Creatinine µmol/L, Low, Week 8, n=282, 275: number analyzed (Participants) | 282 | 275
  Creatinine µmol/L, Low, Week 8, n=282, 275 | 20 | 10
  Creatinine µmol/L, High, Week 8, n=282, 275: number analyzed (Participants) | 282 | 275
  Creatinine µmol/L, High, Week 8, n=282, 275 | 7 | 5
  GGT U/L, Low, Week 4, n=283, 279: number analyzed (Participants) | 283 | 279
  GGT U/L, Low, Week 4, n=283, 279 | 8 | 3
  GGT U/L, High, Week 4, n=283, 279: number analyzed (Participants) | 283 | 279
  GGT U/L, High, Week 4, n=283, 279 | 4 | 3
  GGT U/L, Low, Week 8, n=282, 275: number analyzed (Participants) | 282 | 275
  GGT U/L, Low, Week 8, n=282, 275 | 10 | 6
  GGT U/L, High, Week 8, n=282, 275: number analyzed (Participants) | 282 | 275
  GGT U/L, High, Week 8, n=282, 275 | 4 | 9
  Glucose mmol/L, Low, Week 4, n=283, 279: number analyzed (Participants) | 283 | 279
  Glucose mmol/L, Low, Week 4, n=283, 279 | 17 | 14
  Glucose mmol/L, High, Week 4, n=283, 279: number analyzed (Participants) | 283 | 279
  Glucose mmol/L, High, Week 4, n=283, 279 | 16 | 31
  Glucose mmol/L, Low, Week 8, n=282, 275: number analyzed (Participants) | 282 | 275
  Glucose mmol/L, Low, Week 8, n=282, 275 | 16 | 16
  Glucose mmol/L, High, Week 8, n=282, 275: number analyzed (Participants) | 282 | 275
  Glucose mmol/L, High, Week 8, n=282, 275 | 21 | 12
  Potassium mmol/L, Low, Week 4, n=283, 279: number analyzed (Participants) | 283 | 279
  Potassium mmol/L, Low, Week 4, n=283, 279 | 3 | 2
  Potassium mmol/L, High, Week 4, n=283, 279: number analyzed (Participants) | 283 | 279
  Potassium mmol/L, High, Week 4, n=283, 279 | 1 | 1
  Potassium mmol/L, Low, Week 8, n=282, 275: number analyzed (Participants) | 282 | 275
  Potassium mmol/L, Low, Week 8, n=282, 275 | 1 | 2
  Potassium mmol/L, High, Week 8, n=282, 275: number analyzed (Participants) | 282 | 275
  Potassium mmol/L, High, Week 8, n=282, 275 | 2 | 1
  Magnesium mmol/L, Low, Week 4, n=283, 279: number analyzed (Participants) | 283 | 279
  Magnesium mmol/L, Low, Week 4, n=283, 279 | 0 | 0
  Magnesium mmol/L, High, Week 4, n=283, 279: number analyzed (Participants) | 283 | 279
  Magnesium mmol/L, High, Week 4, n=283, 279 | 0 | 2
  Magnesium mmol/L, Low, Week 8, n=282, 275: number analyzed (Participants) | 282 | 275
  Magnesium mmol/L, Low, Week 8, n=282, 275 | 0 | 1
  Magnesium mmol/L, High, Week 8, n=282, 275: number analyzed (Participants) | 282 | 275
  Magnesium mmol/L, High, Week 8, n=282, 275 | 0 | 0
  Protein g/L, Low, Week 4, n=283, 279: number analyzed (Participants) | 283 | 279
  Protein g/L, Low, Week 4, n=283, 279 | 16 | 17
  Protein g/L, High, Week 4, n=283, 279: number analyzed (Participants) | 283 | 279
  Protein g/L, High, Week 4, n=283, 279 | 1 | 2
  Protein g/L, Low, Week 8, n=282, 275: number analyzed (Participants) | 282 | 275
  Protein g/L, Low, Week 8, n=282, 275 | 16 | 9
  Protein g/L, High, Week 8, n=282, 275: number analyzed (Participants) | 282 | 275
  Protein g/L, High, Week 8, n=282, 275 | 4 | 2
  Sodium mmol/L, Low, Week 4, n=283, 279: number analyzed (Participants) | 283 | 279
  Sodium mmol/L, Low, Week 4, n=283, 279 | 3 | 6
  Sodium mmol/L, High, Week 4, n=283, 279: number analyzed (Participants) | 283 | 279
  Sodium mmol/L, High, Week 4, n=283, 279 | 1 | 1
  Sodium mmol/L, Low, Week 8, n=282, 275: number analyzed (Participants) | 282 | 275
  Sodium mmol/L, Low, Week 8, n=282, 275 | 5 | 6
  Sodium mmol/L, High, Week 8, n=282, 275: number analyzed (Participants) | 282 | 275
  Sodium mmol/L, High, Week 8, n=282, 275 | 2 | 1
  Urate µmol/L, Low, Week 4, n=283, 279: number analyzed (Participants) | 283 | 279
  Urate µmol/L, Low, Week 4, n=283, 279 | 5 | 5
  Urate µmol/L, High, Week 4, n=283, 279: number analyzed (Participants) | 283 | 279
  Urate µmol/L, High, Week 4, n=283, 279 | 4 | 5
  Urate µmol/L, Low, Week 8, n=282, 275: number analyzed (Participants) | 282 | 275
  Urate µmol/L, Low, Week 8, n=282, 275 | 9 | 7
  Urate µmol/L, High, Week 8, n=282, 275: number analyzed (Participants) | 282 | 275
  Urate µmol/L, High, Week 8, n=282, 275 | 4 | 4
  UN mmol/L, Low, Week 4, n=283, 279: number analyzed (Participants) | 283 | 279
  UN mmol/L, Low, Week 4, n=283, 279 | 3 | 4
  UN mmol/L, High, Week 4, n=283, 279: number analyzed (Participants) | 283 | 279
  UN mmol/L, High, Week 4, n=283, 279 | 9 | 7
  UN mmol/L, Low, Week 8, n=282, 275: number analyzed (Participants) | 282 | 275
  UN mmol/L, Low, Week 8, n=282, 275 | 3 | 6
  UN mmol/L, High, Week 8, n=282, 275: number analyzed (Participants) | 282 | 275
  UN mmol/L, High, Week 8, n=282, 275 | 8 | 7

11. Secondary Outcome: Number of Participants With Urinalysis Parameters
Description: Urinalysis parameters included amorphous crystals, bacteria, bilirubin, calcium oxalate (Ca Ox) crystals, choriogonadotropin beta, clarity, color, crystals of Ca Ox, erythrocytes, glucose, hemoglobin, ketone bodies, ketones, leukocyte cell clumps, leukocyte esterase, leukocytes, mucous threads, nitrite, occult blood, protein, specific gravity, squamous epithelial cells, turbidity, urobilinogen, and transitional epithelial cells. In urinalysis test plus sign (+) indicates increase in the level of the parameters.
Time Frame: Day 57
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | AVA Alone | AVA+Raxibacumab
Number analyzed (Participants) | 286 | 280
Participants
  Amorphous crystals 1+ | 1 | 5
  Amorphous crystals 2+ | 7 | 1
  Amorphous crystals 3+ | 0 | 3
  Amorphous crystals 4+ | 3 | 4
  Amorphous crystals trace | 1 | 2
  Bacteria 1+ | 1 | 2
  Bacteria 2+ | 2 | 1
  Bacteria 3+ | 0 | 1
  Bacteria 4+ | 1 | 0
  Bacteria few | 2 | 1
  Bacteria many | 1 | 0
  Bacteria mod | 1 | 2
  Bacteria Occ | 3 | 7
  Bacteria rare | 5 | 8
  Bacteria trace | 2 | 3
  Bilirubin 1+ | 2 | 3
  Bilirubin negative | 196 | 188
  Bilirubin small | 0 | 2
  Ca Ox Crystals few | 0 | 2
  Ca Ox Crystals rare | 2 | 3
  Choriogonadotropin Beta negative | 24 | 16
  Choriogonadotropin Beta positive | 1 | 0
  Clarity, clear | 38 | 44
  Clarity, cloudy | 8 | 2
  Clarity turbid | 1 | 0
  Color amber | 2 | 5
  Color colorless | 1 | 1
  Color light-red | 0 | 1
  Color light-yellow | 6 | 2
  Color yellow | 74 | 71
  Crystals Ca-Ox | 9 | 17
  Erythrocytes 0-2 | 107 | 104
  Erythrocytes 10-25 | 3 | 0
  Erythrocytes 2-5 | 2 | 6
  Erythrocytes 25-50 | 0 | 1
  Erythrocytes 5-10 | 1 | 2
  Erythrocytes 50-99 | 1 | 0
  Erythrocytes innumerable | 0 | 1
  Erythrocytes less than 1 | 10 | 4
  Erythrocytes Tntc | 1 | 0
  Glucose positive | 1 | 0
  Glucose negative | 257 | 257
  Hemoglobin + | 13 | 18
  Hemoglobin ++ | 0 | 3
  Hemoglobin +++ | 1 | 2
  Hemoglobin large | 4 | 2
  Hemoglobin mod | 3 | 6
  Hemoglobin negative | 174 | 166
  Hemoglobin small | 13 | 13
  Hemoglobin trace | 2 | 1
  Ketone bodies negative | 114 | 106
  Ketone bodies trace | 0 | 4
  Ketones + | 1 | 1
  Ketones ++ | 1 | 0
  Ketones ++++ | 0 | 2
  Ketones mod | 1 | 0
  Ketones negative | 255 | 247
  Ketones trace | 0 | 7
  Leukocyte Cell Clumps Occ | 1 | 0
  Leukocyte Cell Clumps rare | 1 | 1
  Leukocyte Esterase 1+ | 4 | 2
  Leukocyte Esterase 2+ | 1 | 1
  Leukocyte Esterase 3+ | 1 | 0
  Leukocyte Esterase large | 10 | 7
  Leukocyte Esterase Mod | 1 | 3
  Leukocyte Esterase Moderate | 1 | 4
  Leukocyte Esterase negative | 162 | 159
  Leukocyte Esterase small | 5 | 7
  Leukocyte Esterase trace | 13 | 10
  Leukocyte + | 5 | 0
  Leukocyte ++ | 1 | 0
  Leukocyte +++ | 1 | 1
  Leukocyte 0-2 | 105 | 99
  Leukocyte 10-25 | 2 | 2
  Leukocyte 2-5 | 6 | 7
  Leukocyte 25-50 | 0 | 1
  Leukocyte 5-10 | 2 | 4
  Leukocyte less than 1 | 8 | 5
  Leukocyte large | 4 | 5
  Leukocyte mod | 1 | 5
  Leukocyte negative | 187 | 188
  Leukocyte small | 2 | 5
  Leukocyte trace | 9 | 7
  Mucous threads 2+ | 0 | 1
  Mucous Threads few | 24 | 25
  Mucous Threads many | 2 | 1
  Mucous Threads Mod | 1 | 2
  Mucous Threads trace | 1 | 2
  Nitrite negative | 190 | 190
  Nitrite positive | 8 | 3
  Occult Blood 1+ | 1 | 0
  Occult Blood 2+ | 1 | 2
  Occult Blood 3+ | 0 | 1
  Occult Blood large | 5 | 3
  Occult Blood mod | 1 | 5
  Occult Blood moderate | 2 | 7
  Occult Blood negative | 163 | 148
  Occult Blood small | 22 | 21
  Occult Blood trace | 3 | 6
  Protein + | 7 | 10
  Protein ++ | 2 | 0
  Protein ++++ | 0 | 1
  Protein 1+ | 3 | 4
  Protein large | 1 | 0
  Protein negative | 244 | 238
  Protein non-heam | 1 | 0
  Protein trace | 12 | 15
  Specific Gravity <=1.005 | 1 | 5
  Specific Gravity >=1.030 | 3 | 6
  Squamous Epithelial Cells 0-2 | 8 | 3
  Squamous Epithelial Cells 2-5 | 2 | 5
  Squamous Epithelial Cells 5-10 | 2 | 2
  Squamous Epithelial Cells <1 | 9 | 8
  Turbidity clear | 15 | 15
  Turbidity cloudy | 2 | 3
  Turbidity hazy | 19 | 16
  Urobilinogen <2.0 | 113 | 111
  Urobilinogen less than 2.0 | 33 | 31
  Urobilinogen normal | 47 | 46
  Transitional Epithelial Cells <1 | 2 | 0

ADVERSE EVENTS:
Time Frame: On-treatment SAEs and non-serious AEs were collected from the start of investigational product until Day 183.
Description: Safety Population
Groups:
- Raxibacumab Only and Discontinued Due to AE During Raxibacumab Infusion: During the study, six of 286 raxibacumab-treated subjects (2.1%) had adverse events (AEs) to raxibacumab that required drug discontinuation, administration of additional medications for mitigation of signs and symptoms, and discontinuation from the study. This new arm is included to capture safety data for these 6 subjects.
- AVA + Raxibacumab With no AE During Raxibacumab Infusion That Led to Discontinuation: Participants administered SC 0.5 mL of AVA doses on Days 1, 15, and 29, with the first AVA dose administered immediately after completion of a single 40 mg/kg, IV infusion of raxibacumab dose (Day 1). Participants were premedicated with 25-50 mg of diphenhydramine up to 1 hour prior to the raxibacumab infusion to reduce the risk of infusion reactions.
Arm/Group | AVA Alone | Raxibacumab Only and Discontinued Due to AE During Raxibacumab Infusion | AVA + Raxibacumab With no AE During Raxibacumab Infusion That Led to Discontinuation
All-Cause Mortality (participants affected / at risk) | 1/286 | 0/6 | 1/280
Serious Adverse Events (participants affected / at risk) | 5/286 | 0/6 | 3/280
Other Adverse Events (participants affected / at risk) | 85/286 | 6/6 | 80/280
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AVA Alone (N=286) | Raxibacumab Only and Discontinued Due to AE During Raxibacumab Infusion (N=6) | AVA + Raxibacumab With no AE During Raxibacumab Infusion That Led to Discontinuation (N=280)
Bile Duct Stone (Hepatobiliary disorders) | 0 | NA | 1
Cholecystitis (Hepatobiliary disorders) | 0 | NA | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | NA | 1
Bronchitis (Infections and infestations) | 0 | NA | 1
Toxicity To Various Agents (Injury, poisoning and procedural complications) | 1 | NA | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | NA | 0
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 2 | NA | 0
Completed Suicide (Psychiatric disorders) | 0 | NA | 1
Suicidal Ideation (Psychiatric disorders) | 1 | NA | 0
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | NA | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | NA | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AVA Alone (N=286) | Raxibacumab Only and Discontinued Due to AE During Raxibacumab Infusion (N=6) | AVA + Raxibacumab With no AE During Raxibacumab Infusion That Led to Discontinuation (N=280)
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 1
Ear Discomfort (Ear and labyrinth disorders) | 1 | 0 | 0
Visual Impairment (Eye disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 6 | 0 | 4
Vomiting (Gastrointestinal disorders) | 2 | 0 | 2
Toothache (Gastrointestinal disorders) | 2 | 0 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 0 | 1
Rectal Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Injection Site Reaction (General disorders) | 18 | 0 | 18
Injection Site Erythema (General disorders) | 11 | 0 | 13
Injection Site Pain (General disorders) | 6 | 0 | 8
Injection Site Swelling (General disorders) | 4 | 0 | 3
Injection Site Pruritus (General disorders) | 4 | 0 | 1
Fatigue (General disorders) | 3 | 0 | 1
Injection Site Nodule (General disorders) | 1 | 0 | 2
Feeling hot (General disorders) | 2 | 0 | 0
Pain (General disorders) | 1 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 1
Asthenia (General disorders) | 1 | 0 | 0
Catheter Site Pain (General disorders) | 0 | 0 | 1
Chest Discomfort (General disorders) | 0 | 0 | 1
Induration (General disorders) | 0 | 0 | 1
Infusion Site Bruising (General disorders) | 0 | 0 | 1
Infusion Site Extravasation (General disorders) | 0 | 0 | 1
Injection Site Mass (General disorders) | 0 | 0 | 1
Injection Site Rash (General disorders) | 0 | 0 | 1
Local Swelling (General disorders) | 1 | 0 | 0
Peripheral Swelling (General disorders) | 1 | 0 | 0
Vaccination Site Reaction (General disorders) | 0 | 0 | 1
Seasonal Allergy (Immune system disorders) | 3 | 0 | 1
Urinary Tract Infection (Infections and infestations) | 6 | 0 | 2
Upper Respiratory Tract Infection (Infections and infestations) | 3 | 0 | 4
Bronchitis (Infections and infestations) | 2 | 0 | 1
Viral Upper Respiratory Tract Infection (Infections and infestations) | 3 | 0 | 0
Influenza (Infections and infestations) | 2 | 0 | 0
Pharyngitis Streptococcal (Infections and infestations) | 2 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 1
Tooth Infection (Infections and infestations) | 2 | 0 | 0
Acute Sinusitis (Infections and infestations) | 0 | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 0 | 1
Furuncle (Infections and infestations) | 0 | 0 | 1
Tonsillitis (Infections and infestations) | 1 | 0 | 0
Tooth Abscess (Infections and infestations) | 1 | 0 | 0
Ligament Sprain (Injury, poisoning and procedural complications) | 1 | 0 | 1
Muscle Strain (Injury, poisoning and procedural complications) | 1 | 0 | 1
Animal Bite (Injury, poisoning and procedural complications) | 0 | 0 | 1
Arthropod Bite (Injury, poisoning and procedural complications) | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Foot Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Infusion Related Reaction (Injury, poisoning and procedural complications) | 0 | 4 | 1
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0
Limb Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 | 0 | 1
Skin Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Upper Limb Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Aspartate Aminotransferase Increased (Investigations) | 1 | 0 | 0
Blood Creatine Phosphokinase Increased (Investigations) | 1 | 0 | 0
Hepatic Enzyme Increased (Investigations) | 1 | 0 | 0
Lymphocyte Count Decreased (Investigations) | 1 | 0 | 0
Neutrophil Count Decreased (Investigations) | 1 | 0 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 3 | 0 | 3
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Muscle Tightnes (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle Fatigue (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 6 | 0 | 9
Presyncope (Nervous system disorders) | 1 | 0 | 3
Nerve Compression (Nervous system disorders) | 1 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0
Loss Of Libido (Psychiatric disorders) | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Dry Throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Throat Tightness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Miliaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus Generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash Erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash Generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 3
Flushing (Vascular disorders) | 1 | 0 | 0
Hot Flush (Vascular disorders) | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-04-25): https://cdn.clinicaltrials.gov/large-docs/55/NCT02339155/Prot_000.pdf
  • Statistical Analysis Plan (2015-04-24): https://cdn.clinicaltrials.gov/large-docs/55/NCT02339155/SAP_001.pdf